CLINICAL TRIAL: NCT02241668
Title: Pilot Study to Assess Accuracy of Time-resolved FLT PET and MR Techniques in Determining Treatment-related Necrosis From Recurrent Glioma
Brief Title: Fluoro-L-Thymidine Positron Emission Tomography (FLT PET) vs. Adv. Magnetic Resonance (MR) Techniques in Recurrent Glioma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to other initiatives
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-0283
Record Dates: First submitted 2014-09-02; First posted 2014-09-16 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Brain Tumor
Keywords: Brain tumor; 3'-Deoxy-3'-18f-Fluorothymidine; Fluoro-L-Thymidine Positron Emission Tomography; FLT PET; Magnetic resonance imaging; MRI
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnetic Resonance Spectroscopy; alovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FLT PET Scan + 3'-Deoxy-3'-18f-Fluorothymidine (Experimental): After a magnetic resonance imaging (MRI) scan of brain performed, an FLT PET scan using 3'-Deoxy-3'-18f-Fluorothymidine solution performed. After solution is injected into a vein, the PET scanner takes pictures of the radioactive solution as it moves through the body and collects at various sites in the body. The entire procedure should last about 60-70 minutes.
  Interventions: Procedure: PET Scan; Drug: 3'-Deoxy-3'-18f-Fluorothymidine

INTERVENTIONS:
Procedure: PET Scan — FLT Pet Scan performed about 60 minutes after 3'-Deoxy-3'-18f-Fluorothymidine solution injected.
  Other Names: Positron Emission Tomography
Drug: 3'-Deoxy-3'-18f-Fluorothymidine — 3'-Deoxy-3'-18f-Fluorothymidine solution injected through a central venous catheter after MRI scan. After solution injected into a vein, PET scanner takes pictures of the radioactive solution as it moves through the body and collects at various sites in the body. Entire procedure should last about 60-70 minutes.

SUMMARY:
The goal of this clinical research study is to learn if using a new imaging solution, 3'-Deoxy-3'-18f-Fluorothymidine, in a positron emission tomography (PET) scan can help doctors determine if your brain lesion is from the tumor returning or the effects of previous treatments.

The results of this imaging scan (called an FLT PET scan) will be compared to the results of a Magnetic Resonance Imaging scan, which you have already had or are scheduled to have outside of this study.

DETAILED DESCRIPTION:
FLT PET Scan:

If you are found to be eligible to take part in this study, you will have an FLT PET scan.

An FLT PET scan uses the 3'-Deoxy-3'-18f-Fluorothymidine solution, which contains a small amount of radioactive material. The radioactive nature of the solution allows the scanner to "see" it in certain places in your body. You will receive the solution by vein through a catheter. A central venous catheter is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form.

After the injection, you will need to rest quietly until it is time for the scan. The amount of rest time may vary, but be prepared to wait for about 60 minutes. During the scan, you will lie flat on your back on a table. After the solution is injected into a vein, the PET scanner takes pictures of the radioactive solution as it moves through the body and collects at various sites in the body. By watching how the solution travels through the body and studying where the solution collects, researchers may be able to learn where the disease is in your body. The entire procedure should last about 60-70 minutes.

You must not eat or drink anything except water for at least 6 hours before the FLT PET scan.

About 2 minutes after the FLT solution is injected, blood (about 10 teaspoons) will be drawn from the catheter. This blood will be drawn to measure how much FLT is in your body and may help the study staff understand the images better.

Length of Study:

After the FLT PET scan is complete, your active participation on this study will be over.

Follow-Up Medical Record Review:

About 30 days after the FLT PET scan, you will be contacted by phone by the study staff to check if you are having any side effects. The phone call should last about 15 minutes.

Your medical records will continue to be reviewed for up to an additional 5 years to learn how you are doing, what other treatments you may have had and how they worked, if you had any new brain problems, or if the tumor came back.

This is an investigational study. The 3'-Deoxy-3'-18f-Fluorothymidine solution is not FDA approved or commercially available. At this time, 3'-Deoxy-3'-18f-Fluorothymidine solution is only being used in research.

Up to 20 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is >/= 18 years old, agrees to participate in the clinical study and to complete all required visits and evaluations. The pediatric population has a different disease profile from the glioma patients we hope to recruit. To reduce heterogeneity in the patient population we will not consider patients younger than 18 for this study.
2. Patient is a candidate for cerebral tumor resection due to an enhancing brain lesion, with history of previous pathologically proven primary brain tumor (WHO grade II-IV diffuse glioma)
3. Patient had diffuse glioma (WHO grade 2 - 4) and as part of their treatment received radiation therapy and Temozolomide (a first-line chemotherapeutic agent).
4. Patient will have subsequently developed an enhancing brain mass greater than 1cm in diameter, at least 6 months after finishing radiation therapy (to differentiate from the more acute treatment related effect of "pseudo-progression").
5. As the predominate means of determining TRN versus recurrent glial tumor at MD Anderson, a brain tumor/ necrosis protocol is ordered as clinically indicated.
6. Patient's clinician based on the clinical and MR information wants to proceed with biopsy or surgical resection within 30 days from when the brain tumor MR protocol was performed. The patient meets with the neurosurgeon and agrees to surgical biopsy or resection.
7. Patient is able to understand and give consent to participation in the study
8. Patient has received as part of their care the Brain Tumor Imaging protocol.
9. Patient agrees to undergo, prior to the procedure, FLT PET at CABI

Exclusion Criteria:

1. The patient is found to have unfavorable anatomy to indicate that stereotactic biopsy/ resection could not be safely performed
2. Claustrophobia that does not readily respond to oral medication
3. Allergy to Fluoro-L-Thymidine
4. Pregnant or lactating (Based on self-reported and clinical care testing with physicians before study participation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Performance of Fluoro-L-Thymidine Positron Emission Tomography (FLT PET) and Perfusion Magnetic Resonance Imaging (MRI) in the Diagnosis of Recurrent High-Grade Glial Tumor | 1 day
  Performance (sensitivity, specificity, negative/ positive predictive values) for MR perfusion and FLT PET made using prior reported values (PEI > 20% 10 and normalized uptake >1.3 17, respectively). Particular attention placed on the location for ROI's and pathology sampling in large heterogenous lesions. Additional, exploratory analysis performed to determine post-hoc optimal cut-off values for classifying glioma vs. necrosis. Logistic regression used to fit a model using a combination of a perfusion values, spectroscopy values, diffusion values, and values from FLT PET.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Rohren, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org